CLINICAL TRIAL: NCT01998776
Title: A Double-blind, Randomized, Placebo Controlled Trial of Misoprostol for Healing of Small Bowel Ulcers in Aspirin Users With Small Bowel Bleeding (MISO-SB Study)
Brief Title: Evaluate Misoprostol for the Healing of Small Bowel Ulcers in Low-dose Aspirin Users Complicated by Small Bowel Bleeding
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Francis KL Chan, Professor, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Diagnostic
Other Study IDs: MISO-SB
Record Dates: First submitted 2013-11-25; First posted 2013-12-02 (Estimated); Last update posted 2019-01-31 (Actual); Status verified 2019-01

CONDITIONS: Ulcer Hemorrhage
Keywords: ulcer
MeSH Terms: conditions — Ulcer | interventions — Misoprostol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Misoprostol (Active Comparator): ASA 100 mg daily + misoprostol 200 four times daily (misoprostol group)
  Interventions: Drug: Misoprostol
- Placebo misoprostol (Placebo Comparator): ASA 100 mg daily + placebo misoprostol four times daily (placebo group)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Misoprostol — Misoprostol 200ug four times daily
  Other Names: Cytotec
  Arms: Misoprostol
Drug: Placebo — Placebo Starch four times daily
  Other Names: Placebo Starch
  Arms: Placebo misoprostol

SUMMARY:
ASA is the most commonly drug used worldwide for prevention of cardiovascular diseases. However, ASA is increasingly recognized as a culprit for small bowel bleeding. Small bowel bleeding is notoriously difficult to diagnose because it is beyond the reach of conventional endoscopy. The advent of wireless, video capsule endoscopy has revolutionized the visualization of small bowel. Capsule endoscopy is a pill that contains a tiny camera for capturing pictures of the small bowel after being swallowed. Currently, capsule endoscopy is a recommended noninvasive approach of identifying the source of small bowel bleeding.

Management of ASA-associated small bowel bleeding is a major clinical challenge since there is not a single effective treatment for small bowel ulcer, and continuation of ASA increases the risk of recurrent small bowel bleeding. However, discontinuation of ASA exposes patients to thrombotic complications. Suppression of prostaglandin synthesis is an important mechanism of ASA-induced small injury. Consistent with this theory, preliminary data from a case series showed that misoprostol, a prostaglandin analog, healed small bowel ulcers in ASA users. However, the efficacy of misoprostol in healing ASA-associated small bowel ulcers has not yet been confirmed by prospective randomized trials.

This double-blind clinical trial tests the hypothesis that misoprostol can heal small bowel ulcers in Aspirin users complicated by small bowel bleeding.

DETAILED DESCRIPTION:
ASA is the most commonly drug used worldwide for prevention of cardiovascular diseases. However, ASA is increasingly recognized as a culprit for small bowel bleeding. The latter condition manifests as overt bleeding (i.e., passing black or bright red stool) or occult blood loss (i.e., normal stool but progressive decrease in hemoglobin level), with normal findings in the stomach and colon. Small bowel bleeding is notoriously difficult to diagnose because it is beyond the reach of conventional endoscopy. The advent of wireless, video capsule endoscopy has revolutionized the visualization of small bowel. Capsule endoscopy is a pill that contains a tiny camera for capturing pictures of the small bowel after being swallowed. Currently, capsule endoscopy is a recommended noninvasive approach of identifying the source of small bowel bleeding.

The problem of small bowel bleeding is increasingly recognized, partly because the use of ASA is rising. In a regional hospital in Hong Kong, we diagnose about 100 cases of ASA-associated small bowel overt bleeding/occult blood loss each year. In a prospective cohort study we found that among ASA users with a history of small bowel bleeding, the risk of recurrent small bowel bleeding is 4 times higher in patients who continued to use ASA than in those who discontinued ASA.

Management of ASA-associated small bowel bleeding is a major clinical challenge for two reasons. First, there is not a single effective treatment for small bowel ulcer. Unlike peptic ulcers, injury to the small bowel is acid-independent. Thus, conventional stomach protective drugs cannot heal or prevent small bowel ulcers in ASA users. Neither can switching to other non-ASA anti-platelet drugs reduce the risk of bleeding. Second, we have shown that continuation of ASA increases the risk of recurrent small bowel bleeding. However, discontinuation of ASA exposes patients to thrombotic complications. Currently, there is no local or international guideline on the management of ASA-associated small bowel bleeding.

Suppression of prostaglandin synthesis is an important mechanism of ASA-induced small injury. Consistent with this theory, preliminary data from a case series showed that misoprostol, a prostaglandin analog, healed small bowel ulcers in ASA users. However, the efficacy of misoprostol in healing ASA-associated small bowel ulcers has not yet been confirmed by prospective randomized trials.

ELIGIBILITY:
Inclusion criteria:

1. Suspected small bowel overt bleeding - melena or hematochezia with normal upper endoscopy and colonoscopy
2. Suspected small bowel occult blood loss - defined as a significant decrease in hemoglobin (≥ 2g/dL), with normal upper endoscopy and colonoscopy, confirmed iron deficiency anemia, and absence of other identifiable causes for hemoglobin decrease (e.g. fluid overload, progressive renal failure, malnutrition, or other hematological disorders such as hemolysis or malignancies)
3. Continuous use of ASA for the duration of the trial
4. Age ≥ 18
5. Written informed consent obtained

Exclusion criteria:

Patients are excluded if they have one or more of the following conditions

1. Increased risk of capsule retention (e.g. Gastric outlet obstruction, bypass surgery, Crohn's disease or suspected small bowel stricture)
2. Abnormal findings on upper endoscopy (e.g. Esophageal varices, grade C or D erosive esophagitis, vascular malformations, ulcer, ≥5 erosions, neoplasms) or colonoscopy (e.g. cancer, polyps > 1cm, inflammatory bowel disease, vascular malformations, bleeding hemorrhoids or diverticular disease)
3. Unable to swallow the video capsule
4. Terminal illness
5. Concomitant use of NSAIDs, sucralfate, rebamepide, anticoagulants, corticosteroids (prednisolone > 7.5mg daily or equivalent), and iron supplement
6. Pregnancy or women of child-bearing age without regular use of contraception

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2013-04; Primary Completion 2018-01-22 (Actual); Study Completion 2018-02 (Actual)

PRIMARY OUTCOMES:
Complete healing of small bowel ulcers | 8 weeks
  The primary outcome is complete healing of small bowel ulcers in 8 weeks

SECONDARY OUTCOMES:
Change in numbers of ulcer/erosions, and hemoglobin level | 8 weeks
  Secondary outcomes include change in the numbers of ulcer/erosions and change in blood hemoglobin level from baseline

CONTACTS AND LOCATIONS:
Overall Officials: Francis KL Chan, MD, Principal Investigator — Chinese University of Hong Kong
Locations (2):
- Prince of Wales Hospital, Hong Kong, China
- Department of Gastroenterology, Osaka City University Graduate School of Medicine, Osaka, Japan

REFERENCES:
- [Derived] Kyaw MH, Otani K, Ching JYL, Higashimori A, Kee KM, Watanabe T, Tse YK, Lee V, Tanigawa T, Cheong PK, Suen BY, Fujiwara Y, Lam K, Arakawa T, Chan FKL. Misoprostol Heals Small Bowel Ulcers in Aspirin Users With Small Bowel Bleeding. Gastroenterology. 2018 Oct;155(4):1090-1097.e1. doi: 10.1053/j.gastro.2018.06.056. Epub 2018 Sep 5. PMID 29966612